CLINICAL TRIAL: NCT00003822
Title: A Phase I and Pharmacokinetic Study of SR-45023A During a 14-Day Treatment Schedule
Brief Title: SR-45023A in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Purpose: Treatment
Other Study IDs: CDR0000066975; ILEX-SR101-A9; ILEX-SR101; UARIZ-HSC-98161; NCI-V99-1532
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2001-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — apomine

INTERVENTIONS:
Drug: apomine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of SR-45023A in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of SR-45023A in patients with locally advanced or metastatic solid tumors that are refractory or for which no standard therapy exists. II. Determine the quantitative toxic effects of SR-45023A in these patients. III. Assess the pharmacokinetic profile of SR-45023A in these patients. IV. Identify the antitumor activity of SR-45023A in these patients.

OUTLINE: This is a dose escalation study. Patients receive oral SR-45023A twice daily for 14 days, followed by 7 days rest. On day 14 of course 1, patients receive only one dose of therapy due to pharmacokinetic sampling. Treatment continues every 21 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of SR-45023A until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. Patients are followed until death.

PROJECTED ACCRUAL: Up to 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed locally advanced or metastatic or solid tumors refractory to standard therapy or for which no standard therapy exists (surgery, radiotherapy, and/or chemotherapy) Measurable or evaluable disease by medical photograph, plain x-ray, CT, MRI, palpation, or serum tumor markers at least 2 times upper limit of normal No asymptomatic brain metastases No leukemia, lymphoma, or multiple myeloma

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-1 Life expectancy: At least 12 weeks Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL No coagulation disorders Hepatic: Bilirubin normal AST and ALT no greater than 3 times upper limit of normal (ULN) (no greater than 5 times ULN if liver involvement) Renal: Creatinine less than 1.5 mg/dL Creatinine clearance at least 45 mL/min Cardiovascular: No cardiac conduction abnormalities Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No active infection No concurrent serious systemic disorders No concurrent or recent (within past 6 months) small bowel obstruction, symptoms of small bowel obstruction, or any other gastrointestinal disease

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy No concurrent filgrastim (G-CSF) Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy and recovered No prior SR-45023A No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal cancer therapy (except contraception, hormone replacement therapy, and corticosteroids) Radiotherapy: See Disease Characteristics Prior radiotherapy allowed to less than 25% of the bone marrow and recovered No prior radiotherapy to the whole pelvis No concurrent radiotherapy Surgery: See Disease Characteristics Other: At least 4 weeks since prior investigational agents No other concurrent investigational agents No concurrent anticoagulation therapy (e.g., Coumadin or heparin) No concurrent digoxin, beta blockers, or calcium channel blockers

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1998-08

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Cancer Center, Tucson, Arizona, United States